CLINICAL TRIAL: NCT01556386
Title: Pharmacogenetic Analysis of Korean Pediatric Patients With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo Seop Ahn, MD. Ph D., Professor, Seoul National University Hospital
Other Study IDs: SNUCH-1202
Record Dates: First submitted 2012-03-08; First posted 2012-03-16 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2013-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; single nucleotide polymorphism
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. Candidate genes exhibit polymorphisms and encodes proteins that are involved in the pharmacokinetics and pharmacodynamics of antileukemic agents
     * Priority was given to polymorphism that were demonstrated to be associated with phenotypes in both clinical and preclinical studies.
     * Candidate genes : CYP3A4*1B, CYPA5*3, GSTM1 deletion, GSTP1 313, GSTT1 deletion, MDR exon 21, MDR exon 26, MTHFR 677, MTHFR 1298, NR3C1 1088, RFC 80, TPMT-1 238, TPMT-1 460, TPMT-1 719, VDR intron 8, VDR FokI, ITPA
  2. Blood sample at complete remission→DNA extraction
  3. Total-Plex (multiplex) PCR amplification
  4. Luminex system analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pharmacogenetic analysis, ALL

SUMMARY:
This study is to find out distribution of genetic polymorphisms and genes related to the chemotherapeutic drugs of ALL.

DETAILED DESCRIPTION:
Cure rate of pediatric ALL dramatically improved over 80%. Resistance to drug and hematologic relapse are remaining problem in ALL treatment. One of the explanations of drug resistance and toxicities is the pharmacogenetic effect. Germline polymorphisms in genes that code for proteins involved in the pharmacokinetics and pharmacodynamics of antileukemic agents are various, and inter-patient variability is the main factor for pharmacogenetic difference. Since multiple chemotherapeutic agents are involved in treating ALL, many genes related to the metabolic pathways of those drugs have an effect on the pharmacokinetics of patients with ALL. In Korea, pharmacogenetic study including multiple genetic loci for pediatric ALL has not been reported.In this study, the distribution of genetic polymorphisms and genes related to antileukemic drugs were analyzed, and their relations to the outcome of treatment and relapse rates were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute lymphoblastic leukemia
* In case of informed consent and assent

Exclusion Criteria:

* Paients or parents refusal

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All the patients with acute lymphoblastic leukemia who was diagnosed and treated in SNUCH.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-06; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To find out distribution of genetic polymorphisms genes related to the pharmacodynamics of the ALL therapy | up to 3 years from diagnosis
  * The distribution of each genetic polymorphism is descriped.
  * The differences in genetic polymorphism between risk groups (high vs. standard) are analyzed using the chi-square test or Fisher's exact test.

SECONDARY OUTCOMES:
To see the ethnic difference of genetic polymorphisms related to the chemotehrapeutic drugs of ALL | whenever after diagnosis and genetic analysis (no time frame needed)
  • The differences in genetic polymorphism between other populations (Korean vs. Western or Japanese) are analyzed using the chi-square test or Fisher's exact test.
To find out relation of genetic polymorphisms and clinical outcome (relapse or survival) | up to 3 years from diagnosis
  - Event-free and overall survival are estimated using Kaplan-Meier analysis, and the survival differences according to different genetic polymorphisms and prognostic variables are analyzed by log-rank test.
To find out risk factors of relapse and death | up to 3 years from diagnosis
  - Multivariate analysis is conducted with Cox proportional hazards regression model to analyze predictive factors. For the multivariate analysis, all significant univariate variables are entered in a stepwise, forward-selection protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea